CLINICAL TRIAL: NCT02042560
Title: Study of Immune Thrombocytopenia Pathogenesis: a Multicenter, Open and Controlled Study.
Brief Title: Study of Immune Thrombocytopenia Pathogenesis:
Acronym: PTI PARI
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: LORCERIE PARI 2010
Record Dates: First submitted 2014-01-17; First posted 2014-01-23 (Estimated); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Primary Immune Thrombocytopenia (ITP)
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Patients with ITP
  Interventions: Other: Blood samples; Other: Spleen samples
- Controls
  Interventions: Other: Blood samples

INTERVENTIONS:
Other: Blood samples
Other: Spleen samples
  Groups: Patients with ITP

SUMMARY:
Immune thrombocytopenia (ITP) is an autoimmune disease characterized by a low platelet count responsible for bleedings. The disease is mostly mediated by antiplatelet antibodies produced by specific B cells. However, T cells are also involved but their role is not completely understood.

The aim of this study is to determine the implication of T cells in the pathogenesis of ITP, notably regulatory T cells (Treg, CD4+CD25highFoxp3+), cytotoxic T cells (CD3+CD8+) and T follicular helper cells (TFH, CD3+CD4+CXCR5+PD-1+ICOS+), in blood and in the spleen of primary ITP patients, compared to healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ITP, defined as thrombocytopenia < 30 G/L, once causes related to infection, medication, systemic auto-immune disease or malignant hemopathy have been ruled out
* persons who have provided written informed consent

Exclusion Criteria:

* persons without national health insurance
* persons under 18 years old
* patients under guardianship
* pregnancy
* subjects suffering from a systemic auto-immune disease, cancer, a progressive infection, or treated with steroids or immunosuppressants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with ITP
Sampling Method: Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2011-05-04 (Actual); Primary Completion 2015-03-12 (Actual); Study Completion 2015-03-12 (Actual)

PRIMARY OUTCOMES:
blood level T cell in ITP patients and in healthy controls | baseline
blood level T cell in ITP patients after treatments | change from baseline at 4 to 8 weeks

SECONDARY OUTCOMES:
blood level splenic T cell in ITP patients and in healthy controls | baseline
frequency of innate immune cells (dendritic cells, monocytes, NK cells…) and their functions in blood and spleens, in patients and in controls | through study completion, an average of 3 years
level of T follicular helper cell | through study completion, an average of 3 years

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHU de Besançon, Besançon
  - CHU de Dijon, Dijon
  - CHU de METZ, Metz